CLINICAL TRIAL: NCT03422120
Title: Human Blood Specimen Collection to Evaluate Immune Cell Function
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: ATGen Canada Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 20160012-01H
Record Dates: First submitted 2018-01-17; First posted 2018-02-05 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-01

CONDITIONS: Colorectal Cancer; Surgery; Perioperative Care
Keywords: Immune Suppression; Natural Killer Cell Mediated Immunity; Natural Killer Cell Cytokine Production; Perioperative/Postoperative Complications
MeSH Terms: conditions — Colorectal Neoplasms; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patient and healthy donor blood was drawn at indicated time points into BD Vacutainer Sodium Heparin coated tubes (~30mL/blood draw) and processed within 4 hrs. 1 mL of whole blood was aliquoted into vacutainer tubes containing PromocoaTM and from the remaining whole blood sample peripheral blood mononuclear cells (PBMCs) were isolated by Ficoll density centrifugation prior to cryopreservation in freezing media (10% DMSO and 90% FBS).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Donors: Healthy patients, without a diagnosis of cancer and age>40. The Natural Killer Cell Activity Assay (NKA) will be measured with a blood test.
  Interventions: Other: Natural Killer Cell Activity Assay
- Colorectal Cancer Surgery Patients: Patients >40 years of age with a histologically confirmed diagnosis of primary colorectal cancer and a planned surgical resection of the primary tumour. The Natural Killer Cell Activity Assay (NKA) will be measured at various perioperative time points with a blood test.
  Interventions: Other: Natural Killer Cell Activity Assay

INTERVENTIONS:
Other: Natural Killer Cell Activity Assay — Subjects had a blood test to measure NK cell activity (NKA) at different time points
  Other Names: NK-Vue

SUMMARY:
Natural killer (NK) cells are leukocytes of the innate immune system and play a central role in the control of cancer metastases. NK cells and other innate immune cells often do not function well in patients with cancer and are also profoundly suppressed after cancer surgery. Dr. Auer's Lab and others have shown that NK cells are critically important in the clearance of tumor metastases and that their impairment can be recovered with immune therapy augmenting the innate immune system. Several studies suggest that cancer patients have depressed NK cell cytotoxicity as compared to healthy controls but that following resection of the cancer, NK cell cytotoxicity returns to normal levels. In this observational study, the investigators will measure NK cell cytotoxicity by the gold standard method (51Cr, a chromium51 release assay) and by a new interferon-ɣ (IFN-ɣ) based assay (NK-Vue™) in healthy humans and colorectal cancer (CRC) surgery patients seen a The Ottawa Hospital. The results of this study will determine if the NK-Vue™ is able to discriminate between healthy human volunteers and newly diagnosed cancer patients and is sufficiently sensitive to detect transient NK cell suppression immediately following surgery.

DETAILED DESCRIPTION:
Rationale:

The purpose of this program is to obtain consent for and to outline the process for collection of fresh blood sample from healthy humans and colorectal cancer patients before and after surgical resection.

Procurement of fresh human blood is required for the following:

* To compare NK cell function, measured by two different assays, in healthy humans and newly diagnosed colorectal cancer patients at the Ottawa Hospital.
* To compare NK cell function, measure by two different assays in colorectal surgery patients preoperatively and at various time points postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have had a recent diagnosis of cancer (any stage) and will be undergoing surgery (cancer group)
* Subjects who are being seen by their physician for other reasons, or healthy volunteers (control group)
* Subjects who provide informed consent to participate in the trial
* Subjects >40 years of age

Exclusion Criteria:

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Inability or unwillingness to sign informed consent form
  * History of active viral or bacterial infection
  * History of prescription use of immunosuppressive drugs within the last six months
  * History of anticancer treatments including radiation or chemotherapy
  * History of autoimmune disorders (rheumatoid arthritis, multiple sclerosis, systemic lupus erythematosus, inflammatory bowel disease including Crohn's disease, Type I diabetes, Guillain-Barré syndrome)
  * Known HIV, Hepatitis B, or Hepatitis C infection
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Natural Killer Cell Activity (NKA) at baseline compared to POD1 in CRC surgery patients | baseline vs. Postoeprative Day (POD) 1
  Measure of NK cell IFN-gamma secretion

SECONDARY OUTCOMES:
Natural Killer Cell Activity (NKA) in healthy donors (HD) as compared to colorectal cancer (CRC) patients (at baseline) | baseline
  Measure of NK cell IFN-gamma secretion

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca C Auer, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided